CLINICAL TRIAL: NCT03755349
Title: COveRs to impRove EsthetiC ouTcome After Surgery for Chronic Subdural hemAtoma by buRr Hole Trepanation (CORRECT-SCAR) - a Single-blinded, Randomized Controlled Trial
Brief Title: Covers to Improve Esthetic Outcome After Surgery for Chronic Subdural Hematoma
Acronym: CORRECT-SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2018-01180
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Hematoma, Subdural, Chronic; Hematoma, Subdural, Intracranial; Haematoma;Subdural;Traumatic
Keywords: Burr hole cover; Chronic subdural hematoma; Trepanation; Aesthetic outcome; Complications; Patient satisfaction; Burr hole plate; Scar; Skin depression
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural, Intracranial; Patient Satisfaction; Cicatrix

STUDY DESIGN:
Intervention Model Description: As the evacuation of a cSDH encompasses trepanation of the skull with 2 burr-holes per side (each one in the frontal and parietal skull region), we will perform the study as follows:
  1. In patients with unilateral cSDH, we will cover either both (intervention group) or none of the burr holes with a burr hole cover (control group).
  2. In patients with bilateral cSDH, we will cover one side with burr hole covers (intervention side), while on the other side no burr hole covers are applied (control side).
Who Masked: Participant
Masking Description: Patients will be blinded for allocation to the study group/side, but surgeons will not be. Patients will not be aware of the study group/side, since the operation takes place under general anesthesia. After surgery, it is not possible to see through the skin, whether or not a burr hole cover has been placed.
  The fact that patients are blinded for the study group allocation will be mentioned in the discharge letter (in order to inform the family physician), and the neurosurgical team of nurses and physicians will also be informed not to "unblind" the patient.
  Unblinding (and revealing a participant's allocated intervention) towards the patient is permissible only if the trial is suspended, prematurely terminated due to security concerns or completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Both burr-holes are covered by burr-hole covers in patients with unilateral cSDH. In patients with bilateral cSDH, both burr-holes of the intervention side are covered by burr-hole covers.
  Interventions: Device: Placement of burr-hole covers
- Control group (Active Comparator): None of the burr-holes are covered by burr-hole covers in patients with unilateral cSDH. In patients with bilateral cSDH, both burr-holes on the control side are left uncovered.
  Interventions: Other: No placement of burr-hole covers

INTERVENTIONS:
Device: Placement of burr-hole covers — Placement of a burr-hole cover (Stryker® UN3 BURR HOLE COVER, 20mm, W/TAB, Item code 53-34520) fixed with 2 screws (Stryker® UNIII AXS SCREWS, SELF-DRILLING, 1.5 x 4MM, Item code 56-15934) on each of two burr-holes
  Other Names: Stryker® UN3 BURR HOLE COVER, 20mm, W/TAB, Item code 53-34520; Stryker® UNIII AXS SCREWS, SELF-DRILLING, 1.5 x 4MM, Item code 56-15934
  Arms: Intervention group
Other: No placement of burr-hole covers — In the control group, none of the burr-holes is covered, representing our current standard of care. In patients with bilateral cSDH, none of the burr-holes on the control side are covered with burr-hole covers.
  Arms: Control group

SUMMARY:
The clinical-functional result after frontal and parietal burr-hole trepanation for the treatment of chronic subdural hematoma (cSDH) is effective with regards to control of the hematoma and regression of symptoms (headache, decreased vigilance and neurological deficits). However, in patients the treatment may leave visible depressions of the scalp, just above the trepanation sites, that typically develop gradually after weeks - months after the procedure. A considerable proportion of patients find this aesthetically, functionally and psychologically disturbing; the skin depressions may even cause pain or interfere with activities of daily living, such as combing, etc.

An effective method would exist to avoid this undesired treatment effect: Before the skin is closed, a permeable titanium burr-hole plate could be attached above the trepanation site in order to prevent the skin from sinking into the bony defect. However, this is rarely done today, likely because there is no evidence that this treatment modification is effective and safe. Moreover, as material is implanted, this causes additional costs.

The primary aim of this study is to evaluate whether the application of burr-hole plates on both the frontal and parietal burr-hole in the context of burr-hole trepanation for the treatment of cSDH can improve patient satisfaction with the aesthetic result of the surgery.

In addition, the study is intended to demonstrate that this additional measure will not result in poorer hematoma control, poorer clinical/neurological outcomes, or additional complications for the patient.

In a prospective, single-blind and controlled approach, we randomize 80 patients with uni- or bilateral cSDH into an intervention group (with burr-hole plates) or into a control group (without burr-hole plates).

The primary end result of the study is the patient's reported satisfaction with the aesthetic outcome of the surgical scar. Secondary results are pain, functionality, neurological status, health-related quality of life, residual hematoma volume, and complications (according to Clavien-Dindo scale; especially re-operation rate for recurring cSDH and infections).

The study corresponds to a modern approach, since today's patients not only expect favorable treatment results for their disease, but the therapy should also avoid permanent undesired side-effects, if possible.

ELIGIBILITY:
Participants fulfilling all of the following inclusion criteria are eligible for the study:

* Patients with first-time cSDH (hypodense, isodense, hyperdense or mixed-type in CT-imaging), scheduled for uni- or bilateral double burr hole trepanation under general anesthesia
* Patient age ≥ 18 years
* Patient non-comatose at time of inclusion (GCS > 8 points)
* Patient able to communicate (in terms of ability to hear, see, speak and understand)

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Patient with recurrent cSDH or previous surgery for cSDH
* Patient with cSDH treated by craniotomy or by single burr hole trepanation
* Patient with cSDH treated in local anesthesia
* Patient unlikely to attend the follow-up (due to reasons of residency, dismal prognosis, etc.)
* Pregnancy
* Known allergy against or incompatibility with Titanium
* Known or suspected non-compliance
* Inability to follow the study procedures, e.g. due to psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the aesthetic result of the scar | 90 days postoperative +/- 10 days
  For the primary outcome, patient satisfaction with the aesthetic results of the scars is determined using a patient-rated outcome measure (PROM), the Aesthetic Numeric Analogue (ANA) scale ranging from 0 (dissatisfied) - 10 (very satisfied). Here, on each side, the frontal and parietal scars are measured separately, and the mean scar satisfaction score per side is built by adding the two values and dividing the sum by two in each patient.

SECONDARY OUTCOMES:
Patient satisfaction with the aesthetic result of the scar | 12 months postoperative +/- 30 days
  Patient satisfaction with the aesthetic results of the scars is determined using the ANA scale ranging from 0 (dissatisfied) - 10 (very satisfied)
Impairment in activities of daily living | 90 days and 12 months postoperative
  Impairment in activities of daily living (ADLs), rated as yes vs. no, with the following options: a) hairdressing, b) combing, c) washing, d) other
Skin depression | 90 days and 12 months postoperative
  Rate of skin depression, rated as yes vs. no
EQ-5D Index | 90 days and 12 months postoperative
  Health-related Quality of Life (HrQoL) - as PROM on the EQ-5D - allowing the calculation of the EQ-5D index that ranges from -0.074 (worst hrQoL) - 1.00 (best hrQoL) using European norms
EQ-5D VAS | 90 days and 12 months postoperative
  HrQoL - as PROM on the EQ-5D - allowing the calculation of the EQ-5D VAS (ranging from 0 (worst hrQoL) - 100 mm (best hrQoL))
Neurological outcome | 90 days postoperative
  Neurological outcome - as physician-rated outcome measure by the NIHSS (ranging from 0 (no neurological deficit) - 42 (severe neurological deficits)), performed by a physician who was trained in the use of the scale (certified)
Disability | 90 days postoperative
  Disability, determined by the mRS (ranging from 0 (no disability) to 6 (dead)

OTHER OUTCOMES:
Home time | 90 days and 12 months postoperative
  Home time, as surrogate marker of disability
Safety Outcome - intraoperative complication | Day of surgery
  Any complication occurring during the surgery
Safety Outcome - postoperative complication | 90 days and 12 months postoperative
  Any deviation from the regular postoperative course will be recorded on the Clavien-Dindo grading scale.
Safety Outcome - hematoma recurrence | 90 days and 12 months postoperative
  Hematoma recurrence per side requiring re-operation
Safety Outcome - local wound infection | 90 days and 12 months postoperative
  Local wound infection requiring surgical revision per side
Radiological Outcome - residual hematoma volume | 90 days postoperative
  Residual hematoma volume in ccm3 will be measured per side on the CT scan routinely performed for clinical patient care
Radiological Outcome - absolute hematoma clearance | 90 days postoperative
  Absolute (in ccm3) hematoma clearance per side will be determined by comparing the pre- and postoperative CT scans
Radiological Outcome - relative hematoma clearance | 90 days postoperative
  Relative (in %) hematoma clearance per side will be determined by comparing the pre- and postoperative CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Martin N Stienen, MD, FEBNS, Principal Investigator — University of Zurich & University Hospital Zurich; Luca Regli, MD, Study Chair — University of Zurich & University Hospital Zurich; Menno R Germans, MD, PhD, Principal Investigator — Universitätsspital Zürich
Locations (1):
- University Hospital Zurich & University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available on reasonable request, once the results are published and if approved by the institutional review board (KEK-ZH).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the results are published.
Access Criteria: IPD will be made available on reasonable request, once the results are published and if approved by the institutional review board (KEK-ZH).

REFERENCES:
- [Background] Vasella F, Akeret K, Smoll NR, Germans MR, Jehli E, Bozinov O, Regli L, Stienen MN; CORRECT SCAR study group. Improving the aesthetic outcome with burr hole cover placement in chronic subdural hematoma evacuation-a retrospective pilot study. Acta Neurochir (Wien). 2018 Nov;160(11):2129-2135. doi: 10.1007/s00701-018-3659-9. Epub 2018 Aug 28. PMID 30155645
- [Background] Velz J, Vasella F, Akeret K, Dias SF, Jehli E, Bozinov O, Regli L, Germans MR, Stienen MN; CORRECT-SCAR study group. Patterns of care: burr-hole cover application for chronic subdural hematoma trepanation. Neurosurg Focus. 2019 Nov 1;47(5):E14. doi: 10.3171/2019.8.FOCUS19245. PMID 31675709
- [Background] Stienen MN, Akeret K, Vasella F, Velz J, Jehli E, Scheffler P, Voglis S, Bichsel O, Smoll NR, Bozinov O, Regli L, Germans MR; CORRECT-SCAR study group*. COveRs to impRove AesthetiC ouTcome after Surgery for Chronic subdural haemAtoma by buRr hole trepanation (CORRECT-SCAR): protocol of a Swiss single-blinded, randomised controlled trial. BMJ Open. 2019 Dec 6;9(12):e031375. doi: 10.1136/bmjopen-2019-031375. PMID 31811007
- [Derived] Stienen MN, Akeret K, Vasella F, Velz J, Jehli E, Voglis S, Bichsel O, Smoll NR, Bozinov O, Regli L, Germans MR; CORRECT-SCAR Study Group. COveRs to impRove EsthetiC ouTcome after Surgery for Chronic subdural hemAtoma by buRr hole trepanation-Results of a Swiss Single-Blinded, Randomized Controlled Trial. Neurosurgery. 2023 Dec 7. doi: 10.1227/neu.0000000000002778. Online ahead of print. PMID 38059611